CLINICAL TRIAL: NCT04084171
Title: Safety of the Tandem t:Slim X2 With Control-IQ Automated Insulin Delivery System in Preschoolers, Age 2-6 Years Old
Brief Title: Safety of Artificial Pancreas Therapy in Preschoolers, Age 2-6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: DexCom, Inc. (Industry); Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Principal Investigator, Marc Breton, Associate Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 190031
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Results first posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Type 1 Diabetes
Keywords: Artificial Pancreas (AP); Continuous Glucose Monitor (CGM); Closed Loop Control (CLC); Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Artificial Pancreas Therapy (Experimental): Subjects will use the Tandem t:slim X2 with Control-IQ Technology + Dexcom G6 to automatically modulate their insulin delivery and control their glycemia.
  Interventions: Device: Tandem t:slim X2 with Control-IQ Technology + Dexcom G6

INTERVENTIONS:
Device: Tandem t:slim X2 with Control-IQ Technology + Dexcom G6 — Subjects will use the Tandem t:slim X2 with Control- IQ Technology and Dexcom G6 CGM to control their glycemia. The Tandem t:slim X2 with Control-IQ device is an automated insulin delivery pump that automatically adjusts insulin delivery to predicted and prevailing glucose levels, as measured by a Dexcom G6 continuous glucose monitor [CGM].
  Other Names: Artificial Pancreas; Automated Insulin Delivery Device

SUMMARY:
A single-arm, multi-center, clinical study to assess the safety profile of the Tandem t:slim X2 with Control-IQ system in children with T1D aged 2-6 years old under free living condition

DETAILED DESCRIPTION:
This clinical trial aims to demonstrate the safety of the Closed-Loop Control (CLC), also known as Artificial Pancreas (AP) named t:slim X2 with Control-IQ Technology and assess usability in a supervised setting for the treatment of type 1 diabetes (T1D) in young children (2-6 years old).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 2 and < 6 years old at the time of consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least 3 months and using insulin at the time of enrollment
3. Use of an insulin pump in the past 3 months
4. Use of Dexcom G6 for at least 11 out of the last 14 days
5. Parent/guardian(s) have familiarity with and use of carbohydrate ratios for meal boluses
6. Living with one or more parent/guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff
7. At least one parent/guardian is willing to stay with the child during the hotel/house portion of the study on the dates selected by the study team
8. Investigator has confidence that the parent/guardian(s) can successfully operate all study devices and is capable of adhering to the protocol
9. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study
10. Total daily insulin dose (TDD) of at least 5 U/day
11. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial
12. Child participant and parent/guardian(s) willingness to participate in all training sessions as directed by study staff
13. Willingness to discontinue non-Tandem t:slim insulin pumps during the entire study
14. Willingness to wear a Dexcom G6 sensor during the entire study
15. An understanding and willingness to follow the protocol and sign informed consent

Exclusion Criteria:

1. Hypoglycemia induced seizure or loss of consciousness in the past 3 months
2. Diabetes Ketoacidosis in the past 3 months
3. Use of diluted insulin
4. Concurrent use of any non-insulin glucose-lowering agent
5. Hemophilia or any other bleeding disorder
6. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk. These conditions may include:

   * Acute illness at the time of the enrollment visit (fever of 101 or higher, vomiting, diarrhea)
   * Addison's disease
   * Diagnosed at less than 1 year of age without positive antibodies
   * Decreased renal function
   * Cystic fibrosis
   * Other chronic conditions, such as an underlying seizure disorder
7. Participation in another pharmaceutical or device trial at the time of enrollment or during the study.
8. Having a family member(s) employed by Tandem Diabetes Care, Inc. or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Breton, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Barbara Davis Center, University of Colorado, Aurora, Colorado
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
To be determined
Supporting Information: Study Protocol
Time Frame: After manuscript publication

REFERENCES:
- [Result] Ekhlaspour L, Schoelwer MJ, Forlenza GP, DeBoer MD, Norlander L, Hsu L, Kingman R, Boranian E, Berget C, Emory E, Buckingham BA, Breton MD, Wadwa RP. Safety and Performance of the Tandem t:slim X2 with Control-IQ Automated Insulin Delivery System in Toddlers and Preschoolers. Diabetes Technol Ther. 2021 May;23(5):384-391. doi: 10.1089/dia.2020.0507. Epub 2020 Dec 8. PMID 33226837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 participants were enrolled across three clinical sites.
Pre-assignment Details: All participants enrolled completed the study.
Period: Overall Study
Arm/Group | Artificial Pancreas Therapy
Started | 12
Baseline | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Diabetes duration [Mean (Standard Deviation); unit: years] | 2.08 (0.89)
HbA1c (%) [Mean (Standard Deviation); unit: percentage] | 7.3 (0.8)
Weight [Mean (Standard Deviation); unit: kg] | 19.3 (3.1)
Total insulin dose [Mean (Standard Deviation); unit: U/(kg*day)] — Total insulin dose U/(kg*day)
  U/(kg*day) | 0.76 (0.14)
Total daily insulin (units) [Mean (Standard Deviation); unit: units] | 14.6 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome
Description: Percentage of subjects with less than 6% time below 70mg/dL and less than 40% time above 180mg/dL.
Time Frame: Baseline results are from the 2-7 day (median of 4 day) use of Open Loop before the hotel admission. AP results are from the 5 day study admission using Control IQ including 48 hours of supervised hotel admission followed by 72 hours at home.
Measure: Number; unit: percentage of subjects
Groups:
- Artificial Pancreas Therapy: Subjects will use the Tandem t:slim X2 with Control-IQ Technology + Dexcom G6 to automatically modulate their insulin delivery and control their glycemia.
  Tandem t:slim X2 with Control-IQ Technology + Dexcom G6: Subjects will use the Tandem t:slim X2 with Control-IQ Technology and Dexcom G6 CGM to control their glycemia. The Tandem t:slim X2 with Control-IQ device is an automated insulin delivery pump that automatically adjusts insulin delivery to predicted and prevailing glucose levels, as measured by a Dexcom G6 continuous glucose monitor [CGM].
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of subjects
  Baseline | 33
  5 days of AP Therapy | 83

2. Secondary Outcome: Below 70 mg/dl.
Description: Percent of time spent below 70 mg/dl.
Time Frame: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of time
  Baseline | 3.7 [1.5 to 6.4]
  5 days of AP Therapy | 3.2 [1.5 to 4.6]

3. Secondary Outcome: Below 60 mg/dl.
Description: Percent of time spent below 60mg/dl.
Time Frame: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of time
  Baseline | 1.6 [0.3 to 2.8]
  5 days of AP Therapy | 0.7 [0.5 to 1.4]

4. Secondary Outcome: Below 54 mg/dl.
Description: Percent of time spent below 54mg/dL.
Time Frame: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of time
  Baseline | 0.6 [0.1 to 1.6]
  5 days of AP Therapy | 0.3 [0.2 to 0.7]

5. Secondary Outcome: Below 50mg/dl.
Description: Percent of time spent below 50mg/dL.
Time Frame: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of time
  Baseline | 0.2 [0.0 to 0.9]
  5 days of AP Therapy | 0.2 [0.1 to 0.3]

6. Secondary Outcome: Above 180 mg/dl.
Description: Percent of time spent above 180mg/dl.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of time
  Baseline | 34.1 (17.3)
  5 days of AP Therapy | 25.7 (12.1)

7. Secondary Outcome: Above 250mg/dl.
Description: Percent of time spent above 250mg/dl.
Time Frame: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of time
  Baseline | 9.7 [6.1 to 19.5]
  5 days of AP Therapy | 4.2 [2.3 to 9]

8. Secondary Outcome: Above 300 mg/dl.
Description: Percent of time spent above 300 mg/dl.
Time Frame: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of time
  Baseline | 3.4 [0.6 to 5.4]
  5 days of AP Therapy | 0.6 [0.1 to 1.6]

9. Secondary Outcome: Between 70-140mg/dl.
Description: Percent of time spent between 70 mg/dl and 140mg/dl.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of time
  Baseline | 41.8 (15.9)
  5 days of AP Therapy | 51.5 (12.8)

10. Secondary Outcome: Between 70-180mg/dl
Description: Percent of time spent between 70 mg/dl and 180mg/dl.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of time
  Baseline | 61.7 (16.1)
  5 days of AP Therapy | 71.3 (12.5)

11. Secondary Outcome: Number of Hypoglycemia Below 70 mg/dL
Description: Number of hypoglycemia events (below 70 mg/dL).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hypoglycemia event
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
hypoglycemia event
  Baseline | 2.13 (1.36)
  5 days of AP Therapy | 1.79 (0.79)

12. Secondary Outcome: Average Number of Treatments.
Description: Average number of carbohydrate treatments per day. Participants were treated with ~16g fast-acting carbohydrates for CGM readings under 80mg/dL during the day and under 70mg/dL overnight (or at higher glycemic thresholds per parent discretion). A repeat treatment was considered if CGM value was<80mg/dL after ~20min. Hypoglycemic treatments could occur at any time per study physician request
Time Frame: The 5 day period of data collection included 48 hours of supervised hotel admission. The remaining 72 hours consisted of at-home Control IQ use under parental supervision and remote study staff monitoring.
Measure: Mean (Inter-Quartile Range); unit: treatments/day
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
treatments/day | 0.8 [0.3 to 1.4]

13. Secondary Outcome: Average of Carbohydrate Treatments (g).
Description: Average amount of carbohydrates (grams) used as a treatment. Participants were treated with ~16g fast-acting carbohydrates for CGM readings under 80mg/dL during the day and under 70mg/dL overnight (or at higher glycemic thresholds per parent discretion). A repeat treatment was considered if CGM value was<80mg/dL after ~20min. Hypoglycemic treatments could occur at any time per study physician request
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
grams | 17.5 (17.6)

14. Secondary Outcome: Percent of Time Spent in Closed Loop
Description: Percentage of the amount of time spent with the Control-IQ system running in closed loop mode.
Time Frame: as for outcome 12
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of time | 96.6 [93.6 to 98.9]

15. Secondary Outcome: CGM Consensus Goal
Description: Percentage of subjects with more than 70% time in 70-180mg/dL range with less than 4% time below 70mg/dL.
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Artificial Pancreas Therapy
Number analyzed (Participants) | 12
percentage of participants
  Baseline | 8
  5 days of AP Therapy | 58

ADVERSE EVENTS:
Time Frame: Up to 14 days
Description: Any untoward medical occurrence in a study participant, irrespective of the relationship between the adverse event and the device(s) under investigation for reportable adverse events for this protocol.
Arm/Group | Artificial Pancreas Therapy
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Short term study in a limited number of individuals significantly limits the generalization of the results to clinical care

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT04084171/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT04084171/ICF_001.pdf